CLINICAL TRIAL: NCT01524068
Title: A Multicenter, Open-Label, Phase II Study of Combined Plasma Exchange (PEX), Rituximab, and Corticosteroids in Patients With Acute Idiopathic Pulmonary Fibrosis Exacerbations
Brief Title: A MultiCenter Study of Combined PEX, Rituximab, and Steroids in Acute Idiopathic Pulmonary Fibrosis Exacerbations
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO12010444
Record Dates: First submitted 2012-01-27; First posted 2012-02-01 (Estimated); Last update posted 2016-01-05 (Estimated); Status verified 2016-01

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Acute Idiopathic Pulmonary Fibrosis Exacerbations; Idiopathic Pulmonary Fibrosis; IPF
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Plasma Exchange; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A - Standard Steroid Treatment (Experimental)
  Interventions: Drug: Standard Steroid Treatment
- Arm B - Experimental Treatment (Experimental)
  Interventions: Drug: The Standard Steroid Treatment, Plasma Exchange and rituximab

INTERVENTIONS:
Drug: Standard Steroid Treatment — One gm of methylprednisolone i.v., on day 0, followed by 40 mg/day i.v. on days 1-4, and days 6-12 (or the p.o. prednisone equivalent). Methylprednisolone 100 mg i.v. will be administered on days 5 and 13. Steroid doses will then be 20 mg methylprednisolone i.v. (or p.o. prednisone equivalent) from days 14-28, and then reduced thereafter at the discretion of the PI at each site.
  Arms: Arm A - Standard Steroid Treatment
Drug: The Standard Steroid Treatment, Plasma Exchange and rituximab — The Standard Steroid Treatment and, after insertion of a dialysis/apheresis catheter into a central vein, followed by initiation of the PEX and rituximab regimens.
  Arms: Arm B - Experimental Treatment

SUMMARY:
This is a randomized, multi-center, open-label Phase II clinical trial to determine the efficacy of combined plasma exchange (PEX), rituximab, and conventional corticosteroid administration, in comparison to corticosteroids alone, among patients with acute Idiopathic Pulmonary Fibrosis (IPF) exacerbations.

The investigators central hypothesis is that antibody-mediated autoimmunity can play an important role in IPF exacerbations. The investigators propose to test our central hypothesis by establishing the efficacy of autoantibody removal by plasma exchange (PEX), in conjunction with B-cell depletion by rituximab to deplete immunoglobulins and minimize their further production, among patients with acute IPF exacerbations.

The primary goal of this randomized, multi-center, open-label Phase II clinical trial is to determine effects of combined plasma exchange (PEX), rituximab, and conventional corticosteroid administration on selected, relevant immunological parameters, in comparison to effects of steroids alone, among AE-IPF patients. The investigators anticipate the findings of this will lead to larger incremental trial(s) to determine actual clinical efficacy of this treatment.

A total of 40 subjects will be enrolled in this multi-center trial from 5 participating medical centers.

DETAILED DESCRIPTION:
This is a randomized, multi-center, open-label Phase II clinical trial to determine the efficacy of combined plasma exchange (PEX), rituximab, and conventional corticosteroid administration, in comparison to corticosteroids alone, among patients with acute IPF exacerbations.

ELIGIBILITY:
INCLUSION CRITERIA:

1. A diagnosis of idiopathic pulmonary fibrosis that fulfills American Thoracic Society Consensus Criteria.1
2. Unexplained worsening or development of dyspnea or hypoxemia within the preceding 30 days.
3. Radiographic imaging showing ground-glass abnormality and/or consolidation superimposed on a reticular or honeycomb pattern consistent with UIP.

EXCLUSION CRITERIA

1. Diagnosis of documented infection, thromboembolic disease, an additional etiology for acute lung injury/adult respiratory distress syndrome, congestive heart failure.
2. Presence of active hepatitis B infection.
3. Coagulopathy defined as an INR > 1.8, PTT > 2 x control, and platelet count < 50K.
4. Hyperosmolar state or diabetic ketoacidosis to suggest uncontrolled diabetes mellitus or uncontrolled hypertension.
5. Hemodynamic instability.
6. History of reaction to blood products, murine-derived products, or prior exposures to human-murine chimeric antibodies,
7. History of malignancy.
8. Unwillingness to accept a blood transfusion.
9. Unwillingness to agree to full supportive medical care (e.g., intubation) for up to 2 weeks after enrollment.
10. Inability or unwillingness to complete post-treatment surveillance for 60 days.
11. Diagnosis of major comorbidities expected to interfere with subjects study participation for 28 days.
12. Treatment for >5 days within the preceding month with >20 mg prednisone (or equivalent dose corticosteroid) or any treatment during the preceding month with a potent cellular immunosuppressant (e.g., cyclophosphamide, methotrexate, mycophenolate, azathiaprine, calcineurin inhibitors, etc.) unless the patient has a BAL negative for opportunistic pathogens (e.g, Pneumocystis, viruses, intracellular organisms, mycobacteria, etc.).
13. Current treatment with an angiotensin converting enzyme inhibitor that cannot be discontinued and/or substituted with another antihypertensive agent (to minimize potential hemodynamic complications during PEX).

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2016-06 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Reduction of autoantibody titers | Baseline to Day 28
  The primary end-point is reduction of autoantibody titers to cultured human primary pulmonary cells, comparing baseline measures of each individual to results of their measures on day 28, or the latest measure among patients who do not survive to day 28.

SECONDARY OUTCOMES:
IgG concentrations | Baseline to Day 60
  Treatment-related effects on plasma IgG concentrations
B-cell counts | Baseline to Day 60
Adverse event (AE) rates | Baseline to Day 60

CONTACTS AND LOCATIONS:
Overall Officials: Steven Duncan, MD, Principal Investigator — University of Pittsburgh
Locations (5):
- United States (5):
  - Geisinger Medical Center, Danville, Pennsylvania
  - Temple University Medical Center, Philladelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Medical Branch - Galveston, Galveston, Texas
  - Inova Fairfax Heart and Vascular Institute, Falls Church, Virginia